CLINICAL TRIAL: NCT02730559
Title: Motivational Interviewing With Dyslipidemic Adolescents Together With a Parent Versus With Adolescents Alone: A Mixed Methods Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Brian McCrindle, Staff Cardiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000035605
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Dyslipidemias
Keywords: Motivational Interviewing
MeSH Terms: conditions — Dyslipidemias | interventions — Motivational Interviewing; Counseling

ARMS (2):
- Intervention Group (Experimental): Group A (Parent-adolescent dyads)
  Interventions: Other: Motivational Interviewing/Counselling
- Control Group - Active Comparator (Active Comparator): Group B (Adolescents only)
  Interventions: Other: Motivational Interviewing/Counselling

INTERVENTIONS:
Other: Motivational Interviewing/Counselling — Motivational Interviewing/Counselling

SUMMARY:
The primary focus of this proposal is to address growing concern of overweight/ obese adolescents with hyperlipidemia. The proposed study is a 2-arm randomized controlled clinical trial to compare the effectiveness of Motivational interviewing (MI) interventions with the parent and adolescent dyad versus adolescent (10-17yr) alone. The patients will be recruited from the Lipid clinic at Sick Kids. The study hypothesis is that parent child dyad will have more success due to the possible synergetic effect compared to adolescents alone. The study's primary outcome is cholesterol levels (Triglycerides/HDL ratio) and secondary outcomes include overall improvement in their lifestyle and their responses to the MI intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age at randomization: 10-17 years old
* 12 hour fasting lipid profile with triglycerides ≥39 mg/dL (1.0 mmol/L) or HDL-C ≤46 mg/dL (1.2 mmol/L), and with non-HDL-C ≥123 mg/dL (3.2 mmol/L)
* Waist to height ratio ≥0.5.

Exclusion Criteria:

* On lipid lowering medication
* non-English speaking
* Developmentally delayed

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in total cholesterol to HDL-C ratio | Initial clinic visit (baseline); Repeated 6 months after baseline;